CLINICAL TRIAL: NCT01805570
Title: Rapid Activity of Platelet Inhibitor Drugs Study (RAPID 2)
Brief Title: Rapid Activity of Platelet Inhibitor Drugs Study 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Antoniucci (Other)
Collaborators: A.R. CARD Onlus Foundation (Other)
Responsible Party: Sponsor-Investigator, David Antoniucci, Head Division of Invasive Cardiology, Careggi Hospital
Organization: Careggi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAPID STUDY 2
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Myocardial Infarction
Keywords: platelet inhibitor; ST-segment Elevation; Myocardial Infarction; stent; prasugrel; ticagrelor
MeSH Terms: conditions — Myocardial Infarction | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel loading dose (Active Comparator): 25 patients with STEMI undergoing PPCI with bivalirudin (GP IIb/IIIa not allowed) will be randomized to receive Prasugrel before PPCI.
  Interventions: Drug: Prasugrel
- Ticagrelor loading dose (Active Comparator): 25 patients with STEMI undergoing PPCI with bivalirudin (GP IIb/IIIa not allowed) will be randomized to receive Ticagrelor before PPCI.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — 25 patients with STEMI undergoing PPCI with bivalirudin (GP IIb/IIIa not allowed) will be randomized to receive Prasugrel before PPCI. The loading dose of Prasugrel will be 60 mg. The loading dose will be performed as soon as possible in the Emergency Room or in the Cath Lab. In the case of vomit in the first hour after drug loading dose a new reduced loading dose will be administered .
  Arms: Prasugrel loading dose
Drug: Ticagrelor — 25 patients with STEMI undergoing PPCI with bivalirudin (GP IIb/IIIa not allowed) will be randomized to receive Ticagrelor before PPCI. The loading dose of Ticagrelor will be 360 mg. The loading dose will be performed as soon as possible in the Emergency Room or in the Cath Lab. In the case of vomit in the first hour after drug loading dose a new reduced loading dose will be administered .
  Arms: Ticagrelor loading dose

SUMMARY:
The aim of the RAPID study is to evaluate the superiority rapid onset of action of Ticagrelor 360 mg LD versus Prasugrel 60 mg LD, in 50 patients with STEMI (ST segment elevation myocardial infarction) undergoing PPCI with bivalirudin monotherapy. Secondary study aim is to found out clinical predictors of high residual platelet reactivity in the first hour after a novel oral antiplatelet agent LD.

DETAILED DESCRIPTION:
50 consecutive patients with STEMI undergoing PPCI with bivalirudin (GP IIb/IIIa not allowed) will be randomized to receive Prasugrel (n= 25) or Ticagrelor (n= 25) before PPCI ( primary percutaneous coronary intervention) in a open label fashion. The loading dose of Prasugrel will be 60 mg, the loading dose of Ticagrelor will be 360 mg in 25 patients. The loading dose will be performed as soon as possible in the Emergency Room or in the Cath Lab. In the case of vomit in the first hour after drug loading dose a new reduced loading dose will be administered (30 mg Prasugrel or 180 mg Ticagrelor). All interventions will be performed by the femoral approach according to current standards. The use of thrombectomy before infarct-related artery stenting, of everolimus eluting stent and of closure devices will be strongly encouraged. Bivalirudin will be administered as a bolus 0.75 mg/kg followed by 1.75 mg/kg/h infusion during PCI. After PCI (percutaneous coronary intervention) a reduced bivalirudin infusion of 0.25 mg/kg/h for 4 hours will be allowed. Dual antiplatelet therapy (100 mg aspirin associated with 5 or 10 mg Prasugrel or 180 mg Ticagrelor) will be recommended for 12 months.

Residual platelet reactivity will be assessed in all patients at baseline (time of LD), and after 1, 2, 4 and 12 hours by a point-of-care test VerifyNow bedside available in the Intensive cardiac care Unit. High residual platelet reactivity will be defined as a Platelet Reactivity Units (PRU) > 240 by VerifyNow. At the same time point, Aspirin Reactivity Units (ARU) by VerifyNow will be also assessed. Follow-up will be performed by outpatient visits or telephone interviews at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting within 12 hours from the onset of symptoms with STEMI (ST segment elevation myocardial infarction)
* Informed, written consent

Exclusion Criteria:

* Age < 18 years or Age > 75 years
* Active bleeding; bleeding diathesis; coagulopathy
* Increased risk of bradycardiac events
* History of gastrointestinal or genitourinary bleeding <2 months
* Major surgery in the last 6 weeks
* History of intracranial bleeding or structural abnormalities
* Suspected aortic dissection
* Any previous TIA (transient ischemic attack)/stroke
* Any other condition that may put the patient at risk or influence study results or investigator's opinion (severe haemodynamic instability, known malignancies or other comorbid conditions with life expectancy <1 year)
* Administration in the week before the index event of clopidogrel, ticlopidine, prasugrel, ticagrelor, thrombolytics, bivalirudin, low-molecular weight heparin or fondaparinux .
* Concomitant oral or IV therapy with strong CYP3A inhibitors or strong CYP3A inducers, CYP3A with narrow therapeutic windows
* Known relevant hematological deviations: Hb <10 g/dl, Platelet count <100x10^9/l
* Use of coumadin derivatives within the last 7 days
* Chronic therapy with prasugrel or ticagrelor
* Known severe liver disease, severe renal failure
* Known allergy to the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Residual Platelet Reactivity by VerifyNow | 1 hour
  residual platelet reactivity by Platelet Reactivity Units (PRU) VerifyNow 1 hour after oral antiplatelet agent LD.

SECONDARY OUTCOMES:
High residual platelet reactivity | 2,4,12 hours
  High residual platelet reactivity will be defined as a Platelet Reactivity Units (PRU) > 240 by VerifyNow

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Principal Investigator — Careggi Hospital, Division of Invasive Cardiology
Locations (1):
- Careggi Hospital, Florence, Italy

REFERENCES:
- [Derived] Parodi G, Bellandi B, Valenti R, Migliorini A, Marcucci R, Carrabba N, Giurlani L, Gensini GF, Abbate R, Antoniucci D. Comparison of double (360 mg) ticagrelor loading dose with standard (60 mg) prasugrel loading dose in ST-elevation myocardial infarction patients: the Rapid Activity of Platelet Inhibitor Drugs (RAPID) primary PCI 2 study. Am Heart J. 2014 Jun;167(6):909-14. doi: 10.1016/j.ahj.2014.03.011. Epub 2014 Apr 4. PMID 24890542